CLINICAL TRIAL: NCT03160235
Title: Development of MRI Protocols and Associated Explorations (EEG, NIRS) in Voluntary Patients
Acronym: MAP-PV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC12.239
Record Dates: First submitted 2017-04-24; First posted 2017-05-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Electroencephalography

STUDY DESIGN:
Intervention Model Description: Methodological development of new MRI approaches
Masking Description: Magnetic resonance imaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Development of MRI protocols (Experimental): MRI exam to grade differents interventions for future research
  Interventions: Radiation: Magnetic resonance imaging
- Development of EEG protocols (Experimental): EEF exam to grade differents interventions for future research
  Interventions: Device: EEG
- Development of NIRS protocols (Experimental): NIRS exam to grade differents interventions for future research
  Interventions: Device: NIRS

INTERVENTIONS:
Radiation: Magnetic resonance imaging
  Arms: Development of MRI protocols
Device: EEG
  Arms: Development of EEG protocols
Device: NIRS
  Arms: Development of NIRS protocols

SUMMARY:
Studies that will be carried out on healthy volunteers will have as main objective the development and optimization of the parameters of sequences or the design of the paradigms of stimulation in order to optimize the quality and the relevance of the images realized taking in Taking account of anatomical, functional or metabolic parameters, or integrating new approaches resulting from technical evolutions

DETAILED DESCRIPTION:
The pathologies that interest us in these refinements concern mainly the chronic (or sequellar) brain disorders which can be degenerative, developmental or vascular. The patients who will be recruited will be known patients of our Service (University Clinic of Neuroradiology and MRI) that we follow during checks. The type of examination that will be applied to them, between MRI, EEG and NIRS, will be specified in the consent form. These examinations will not be invoiced either to the patient or to the social security, and the related costs will be borne by our Federative Research Structure or sometimes, when these explorations are upstream of a defined research protocol and funded, They will be financed under this protocol.

ELIGIBILITY:
Inclusion Criteria:

* major voluntary patients
* socially insured.
* Karnofsky score above 60%.
* given their consent.
* absence of contraindication to the MRI examination

Exclusion Criteria:

* Subjects under the age of 18
* pregnant women
* persons referred to in articles L1121-5 to L1121-8 of the CSP.
* Patients with acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Spatial resolution of new MRI imaging sequences MRI scanning. | Two hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No